CLINICAL TRIAL: NCT03586245
Title: Iron Absorption From Iron Enriched Aspergillus Oryzae in Females Using Stable Iron Isotope Methodology.
Brief Title: Iron Absorption From Iron Enriched Aspergillus Oryzae in Females Using Stable Isotope Methodology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, Dr. Manju B. Reddy, Professor, Iowa State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ASP Study
Record Dates: First submitted 2018-07-06; First posted 2018-07-13 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2016-08

CONDITIONS: Iron Absorption
Keywords: Iron Bioavailability; Iron Fortification; ferrous sulfate; ferric pyrophosphate; aspergillus oryzae; stable isotope
MeSH Terms: interventions — ferric pyrophosphate; ferrous sulfate

STUDY DESIGN:
Intervention Model Description: Subjects consumed two stable isotopes (57Fe and 58Fe). Study I, three consecutive days of meal A followed by crossover of three days meal B were consumed. Study II was a crossover between meal B and meal C.
Who Masked: Participant
Masking Description: All stable isotopes (FePP, ASP, FeSO4) were all individually added to test meal and mixed thoroughly by investigators. Participants were brought the meal to consume, unknowingly of which respective treatment they were receiving.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ferric pyrophosphate (Active Comparator): Study I group was required to consume a total of 3 meals. Each meal contained 4.2 mg added iron compounds.
  * 57FePP (95.8%) 3.49 mg
  * Aspergillus oryzae (unenriched) 0.025 mg
  * FePP natural abundance 0.685 mg.
  Subjects received iron fortificants in a meal composed of zucchini, cabbage, carrot (42g each), onion (24g), corn oil (6.3 g), jasmine rice (75g dw), and flavored granulated chicken bouillon (6.6g). All meals were consumed in a fasted state with nothing to eat or drink (besides water) for 3 hours following consumption.
  Interventions: Dietary Supplement: Ferric pyrophosphate
- Aspiron (Experimental): The Aspiron group was required to follow the same protocol as the 57Fe as FePP, with the exception of consuming 58Fe ASP.
  * ASP-p (8% Fe; natural abundance) 3.516 mg
  * 58ASP-p (5% Fe; 99.5% enrichment) 0.68 mg
  * 4.2 total mg of Fe
  Interventions: Dietary Supplement: Aspiron
- Ferrous sulfate (Other): The FeSO4 study group was required to consume a total of 3 meals. Each meal contained 4.2 mg added iron compounds. .
  * Aspergillus oryzae (unenriched) 0.027 mg
  * 57FeSO4 (95.4%) 3.18 mg
  * 4.2 total mg of Fe
  Interventions: Dietary Supplement: Ferrous sulfate

INTERVENTIONS:
Dietary Supplement: Ferric pyrophosphate — 57 Iron isotopically labeled FePP powder.
  Arms: Ferric pyrophosphate
Dietary Supplement: Aspiron — 58 Iron isotope intrinsically labeled Aspergillus oryzae.
  Arms: Aspiron
Dietary Supplement: Ferrous sulfate — 57 Iron isotopically labeled FeSO4 powder.
  Arms: Ferrous sulfate

SUMMARY:
The objective of this study was to compare the iron absorption from ferric pyrophosphate enriched Aspergillus oryzae (ASP-p) to commonly used ferric pyrophosphate (FePP) and ferrous sulfate (FeSO4) when fortified in chicken bouillon, using stable isotope methodology.

DETAILED DESCRIPTION:
Iron deficiency anemia (IDA) remains the most common nutrient deficiency, globally. Consequences such as decreased cognition, growth impairment, and morbidity and mortality arise from inadequate iron intake. Many technological challenges are presented in fortifying foods with iron, as inorganic iron salts are known to cause organoleptic problems in the food. As a result, finding an iron fortificant that doesn't alter taste, smell or stability of the food is ideal, however most suitable iron fortificants contain low bioavailability. Thirty-five non-anemic female subjects with ferritin ≤ 40 µg/L were recruited for both studies (17 in study I; 18 in study II). In both studies, each meal contained a total of 4.2 mg of added iron fortificants to a test meal containing 6.6 g of chicken bouillon. Participants were randomized to consume either meal A or B, followed by B or C. In study I, subjects consumed a total of 10 mg 57Fe as FePP and 2 mg 58Fe as ASP-p each over three consecutive days. Study II, subjects consumed a total of 10 mg 57Fe as FeSO4 and 2 mg 58Fe as ASP-p over 2 weekends. Blood samples collected at baseline were used to measure iron status indicators such as serum ferritin, C-reactive protein, hepcidin and hematocrit. Fourteen days following final isotope dosing, whole blood samples were collected and the fractional iron absorption of each iron fortificant containing labelled stable isotopes was measured via thermal ionization mass spectrometry with estimation of 80% incorporation into the hemoglobin.

ELIGIBILITY:
Inclusion Criteria:

* Suboptimal iron stores (Serum ferritin < 40 µg/L)
* BMI in range 18.5 - 24.9 kg/m2
* Willing to consumed meals containing iron supplement
* Willing to discontinue blood donation two weeks prior and during the study
* Willing to discontinue vitamin and mineral supplement use during the study
* Willing to provide a 15 ml blood for initial screening and 30 ml blood during the study (15 ml at each visit for 2 times in 24 days)
* Willing to attend 8 lab visits during the study

Exclusion Criteria:

* Pregnant
* Lactating
* Smoker
* Anemic (hemoglobin < 120 g/L)
* Has gastrointestinal disease/condition that can affect absorption
* Vegetarian
* Allergic to corn, wheat, soybean nor fungal supplements

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2016-10-28 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Percentage Fractional Iron absorption of FePP, FeS)4 and ASP | Whole blood collected 14 days following isotope consumption to allow for enrichment.
  Isotope enrichment in the whole blood samples after 14 days of feeding the meals assuming 80% incorporation of iron into the hemoglobin. Circulating iron was calculated from blood volume, height (cm), weight (kg) and hemoglobin (g/dL).

CONTACTS AND LOCATIONS:
Overall Officials: Manju B Reddy, PhD, Principal Investigator — Iowa State University

IPD SHARING:
Plan to Share IPD: No
Publish results in a journal.

REFERENCES:
- [Derived] Bries AE, Hurrell RF, Reddy MB. Iron Absorption from Bouillon Fortified with Iron-Enriched Aspergillus oryzae Is Higher Than That Fortified with Ferric Pyrophosphate in Young Women. J Nutr. 2020 May 1;150(5):1109-1115. doi: 10.1093/jn/nxaa035. PMID 32073619